CLINICAL TRIAL: NCT04347746
Title: Comparison of Interventions in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: sg01
Record Dates: First submitted 2020-02-19; First posted 2020-04-15 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Carpal Tunnel Syndrome; Carpal Tunnel Syndrome Bilateral
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical group (Active Comparator): Individuals with bilateral idiopathic CTS with clinical criteria and mild to moderate ENMG severity and symptom evolution time above six months.
  Interventions: Behavioral: stretching physiotherapy; Behavioral: Myofascial therapy
- Surgical group (Active Comparator): Individuals with bilateral idiopathic CTS with clinical criteria and severe ENMG in at least one hand and symptom evolution time above six months. These will be submitted to surgery on the severe hand and if equal severity on both hands, the dominant hand will be operated, with the patient's consent.
  Interventions: Behavioral: stretching physiotherapy; Behavioral: Myofascial therapy

INTERVENTIONS:
Behavioral: stretching physiotherapy — A booklet with images and a description of all movements to be performed during therapy will be offered to patients. The booklet illustrates the movements for stretching the upper limbs divided as follows: three movements for the neck, three movements for the arms and forearms and four movements for the hands.
  The therapy will be carried out twice a week at the Unopar research center, under the guidance of a physiotherapist trained in technique and supervision by a senior therapist. At the end of each movement, the individual is instructed to maintain the position for 40 seconds.
  Patients will be instructed to appear in comfortable clothes and the environment will have favorable conditions.
Behavioral: Myofascial therapy — Myofascial therapy will be performed on the upper limbs, pectoral and dorsal regions with the aid of hooks (instrument assisted soft-tissue mobilization). In the supine position, the pectoral muscles will be manipulated (infracromial, external, axillary-claviculopectoral fossa), biceps brachii (short head, long and forearm insertion), round pronator, anterior forearm musculature (compartment of the radial extensor of the long carpus and brevis, finger extensor and ulnar carpal extensor). In lateral decubitus the deltoid muscle in the anterior, middle and posterior portions. In the prone position, the trapezius muscle (in its cervical, scapular and nuchal insertions), scapular levator muscle, great dorsal muscle (in its lateral insertions) and triceps brachii muscle. The hook manipulation time is two minutes of execution for each muscle mentioned above, making a total time of each section of forty minutes. There will be two weekly sessions with an interval between forty-eight hours.

SUMMARY:
This study aims to compare two types of intervention (stretching and myofascial manipulation) in the treatment of individuals with bilateral idiopathic carpal tunnel syndrome. This comparison applies to two groups, the clinical group is composed of patients of mild or moderate degree, whereas the surgical group is composed of a patient with at least one hand in severe degree and interventions are made after surgery.

DETAILED DESCRIPTION:
Using clinical criteria and ENMG, individuals will be divided into a clinical group when they have a mild and / or moderate degree of involvement in the hands and a surgical group when the impairment intensity is severe in at least one hand.

The individuals in the clinical group will be randomized into two groups, with one group starting with stretching and a second group starting with hook-assisted myofascial manipulation. After four weeks of initial therapy and one week of wash-out the assessment tests described above will be applied. The groups will be inverted, maintaining the duration and frequency of the previous stage of the proposed therapies. After four weeks with a week of wash-out the tests will be reapplied in order to evaluate the therapeutic response.

Individuals with severe idiopathic CTS will undergo surgery using a standard open technique with local anesthesia and after four weeks, randomization will be made for postoperative treatment on both hands by stretching or myofascial manipulation in the same manner described for the clinical group.

Questionnaires will be applied in order to understand the patient's symptoms, functions, pain and quality of life. In addition, tests will be used to assess hand strength, sensitivity and hand ability.

ELIGIBILITY:
Inclusion Criteria:

* bilateral idiopathic CTS above six months of symptomatology;
* with clinical criteria and ENMG for indication of clinical or surgical treatment;
* who have no history of gabapentin allergy.

Exclusion Criteria:

* Individuals with CTS for other reasons, such as pregnancy, arthritis, hypothyroidism, diabetes mellitus, trauma, expansive tunnel damage, amyloids, sarcoidosis, multiple myeloma, and leukemia.
* Individuals with conditions that can simulate CTS, such as carpometacarpal thumb arthritis, cervical radiculopathy mainly of the sixth cervical root level, radial flexor carpal tenosynovitis and central disorders such as multiple sclerosis and cerebral infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline Visual analog scale at eight weeks | Change from baseline at 8 weeks
  The visual analog scale will measure the patient's pain intensity. The scale goes from 0 to 10, with 10 being better.
Change from baseline Boston Questionnarie score at eight weeks | Change from baseline at 8 weeks
  The Boston questionnaire assesses the symptoms and functions of patients with CTS, it is self-administered. The sensitivity scale goes from 11 to 55, the motor scale goes from 7 to 35, bigger is better.

SECONDARY OUTCOMES:
Change from baseline Short-Form 6 Dimensions at eight weeks | Change from baseline at 8 weeks
  The Short-Form 6 Dimensions (SF6) questionnaire will be used to measure the impact on global health status. The scale goes from 0 to 100, with 100 being better.
Change from baseline Hand strength test at eight weeks | Change from baseline at 8 weeks.
  The hand strength test will use the Jammar hydraulic handgrip diameter and the hydraulic Pinch Gauge Jamar hydraulic will be used to measure the force of the digital clamp and digital clamp.
Change from baseline Sensitivity tests at eigth weeks | Change from baseline at 8 weeks
  The sensitivity tests will be evaluated with the Semmes-Weistein monofilaments on the distal digital pulp of the second and fifth fingers, the two-point discriminator Touch-Test on the distal digital pulp of the second and fifth fingers and the vibratory sensitivity with 30 and 259 hertz tuning fork over the distal interphalangeal joint of the second and fifth fingers.
Change from baseline Manual skill score at eigth weeks | Change from baseline at 8 weeks
  Manual skill will be analyzed with the nine-pin box and manual skill panel
Change from baseline Brief Michigan Hand Questionnaire for the right and left hand at eight weeks. | Change from baseline at 8 weeks
  The BMHQ 12 items is an efficient and versatile result instrument, specific to manual disability and the quality of the therapeutic care employed. In addition, this questionnaire retains the psychometric properties of the original MHQ. The scale goes from 0 to 100, with 100 being better.
3D Assessment of Hand Function for the right and left hand. | Day 0
  3D assessement evaluates the hand in relation to pain, its function and its appearance from the perspective of the individual at the expense of the evaluation from the doctor's point of view.

CONTACTS AND LOCATIONS:
Locations (1):
- Unopar, Londrina, Paraná, Brazil